CLINICAL TRIAL: NCT00279695
Title: Ultrasonic Evaluation of Ocular Tissues
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Riverside Research Institute (Other)
Responsible Party: D. Jackson Coleman, MD, Weill Cornell Medical College
Other Study IDs: EB00238; 0703009082
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Glaucoma; Tumors; Age-Related Macular Degeneration
Keywords: Glaucoma; Accommodation; Ocular Tumors; Age-Related Macular Degeneration; Ultrasound; Eye
MeSH Terms: conditions — Glaucoma; Neoplasms; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Subjects with glaucoma and age-matched normals
  Interventions: Procedure: high frequency ultrasound examination
- 2: normal volunteers, two age groups, one 18-25 years old, one 50 years and older.
  Interventions: Procedure: high frequency ultrasound examination
- 3: subjects with tumors of the iris and ciliary body
  Interventions: Procedure: high frequency ultrasound examination
- 4: subjects with age-related macular degeneration and age-matched normals
  Interventions: Procedure: high frequency ultrasound examination

INTERVENTIONS:
Procedure: high frequency ultrasound examination — high frequency ultrasound examination of the eye

SUMMARY:
The objective of this research program is to improve diagnosis and treatment monitoring of ophthalmic disease by improving diagnostic ultrasound techniques. The program explores the use of novel signal and imaging processing techniques towards this end.

DETAILED DESCRIPTION:
This study involves the diagnosis of several eye diseases, as follows:

Glaucoma:

1. Morphometry and spectral parameter assays: Clinical correlative studies in primary and secondary glaucoma subgroups: This is a volunteer study to obtain volumetric measurements of age-related changes in the ciliary body and individual ciliary muscle components. The study will provide baseline values for treatment monitoring studies of glaucoma therapeutics. There is minimal risk that the ultrasound procedure may reveal an occult ocular disease process, but the probability is very small. Patients will be informed and assisted in obtaining appropriate care if any abnormality is seen.
2. Morphometry and spectral parameter assays: Ciliary body drug interactions in patients with initial diagnosis of open angle glaucoma: This study will attempt to document changes in anterior segment functional anatomy related to medical management of glaucoma. We hypothesize that several classes of anti-glaucoma drugs produce permanent modification of ciliary muscle vasculature that is related in turn to loss of drug efficacy over time. Data from COAG patients will be compared with age and sex matched normals. Participation in the study will not effect the ongoing glaucoma therapy of patients.

   Accommodation:
3. Accommodative function in young emmetropes and transitional presbyopes: This is a volunteer study to develop a descriptive model of the human eye's focusing mechanism based on ultrasound morphometric measurements and spectral parameter assays. This study will measure dynamic changes in ciliary body spectral assays (size, CQ2) during calibrated accommodative tasks in volunteers with good amplitude of accommodation and those with accommodative loss do to aging and model 3-D conformal changes in anterior segment structures during accommodation. There is minimal risk that the ultrasound procedure may reveal an occult ocular disease process, but the probability is very small. Patients will be informed and assisted in obtaining appropriate care if any abnormality is seen.

   Ocular Tumors
4. Tumors of the iris and ciliary body: This is an observational study of growth pattern changes in anterior melanoma for the purpose of identifying prognostic variables associated with rapid tumor growth. A percentage of small melanomas are observed for periods of up to several years before demonstrable growth will suggest more aggressive treatment. In the clinical ultrasound practice many patients with these tumors are seen at 3 to 6 month intervals to provide the ophthalmic oncologist with updated tumor volume data. We will examine changes in the ultrasound scattering structure of these tumors over time and their correlation with volume changes. The on-going research data are not released as part of the clinical ultrasound report.

   Age-related Macular Degeneration
5. Posterior examinations: age-related macular degeneration: This study will examine the use of higher frequency (20-30 MHz) ultrasound in the early diagnosis of Age-related macular degeneration. Our hypothesis is that early changes in the choriocapillaries and choroid vascular density and conformation can be detected with high-frequency spectral assays. We will obtain ultrasound scans at frequencies of 20 MHz or more, as well as OCT and fundus photographs. Similar numbers of age-matched control subjects will be examined. Measurements of retinal and choroidal thickness profiles in the peri-macular region will be made. Spectral data will be used for morphologic vascular analysis (size and shape). Statistical comparison will be made using parametric and non-parametric methods between control and AMD groups.

ELIGIBILITY:
Inclusion Criteria:

Have one of the following eye diseases Glaucoma Ocular Tumors Age-Related Macular Degeneration

Exclusion Criteria:

none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ophthalmology practice referrals
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 1996-01; Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: D. Jackson Coleman, MD, Principal Investigator — Weill Cornell Medical College - New York Presbyterian Hospital
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Background] Silverman RH, Ursea R, Kruse D, Ferrara KW, Rondeau MJ, Coleman DJ. Ultrasound measurement of the effect of temperature on microperfusion in the eye. Ultrasound Med Biol. 2002 Nov-Dec;28(11-12):1413-9. doi: 10.1016/s0301-5629(02)00694-4. PMID 12498936
- [Background] Silverman RH, Kruse DE, Coleman DJ, Ferrara KW. High-resolution ultrasonic imaging of blood flow in the anterior segment of the eye. Invest Ophthalmol Vis Sci. 1999 Jun;40(7):1373-81. PMID 10359319
- [Result] Rondeau MJ, Barcsay G, Silverman RH, Reinstein DZ, Krishnamurthy R, Chabi A, Du T, Coleman DJ. Very high frequency ultrasound biometry of the anterior and posterior chamber diameter. J Refract Surg. 2004 Sep-Oct;20(5):454-64. doi: 10.3928/1081-597X-20040901-08. PMID 15523957
- [Result] Coleman DJ, Silverman RH, Chabi A, Rondeau MJ, Shung KK, Cannata J, Lincoff H. High-resolution ultrasonic imaging of the posterior segment. Ophthalmology. 2004 Jul;111(7):1344-51. doi: 10.1016/j.ophtha.2003.10.029. PMID 15234135
- [Result] Coleman DJ, Silverman RH, Rondeau MJ, Boldt HC, Lloyd HO, Lizzi FL, Weingeist TA, Chen X, Vangveeravong S, Folberg R. Noninvasive in vivo detection of prognostic indicators for high-risk uveal melanoma: ultrasound parameter imaging. Ophthalmology. 2004 Mar;111(3):558-64. doi: 10.1016/j.ophtha.2003.06.021. PMID 15019336
- [Result] Silverman RH, Folberg R, Rondeau MJ, Boldt HC, Lloyd HO, Chen X, Lizzi FL, Weingeist TA, Coleman DJ. Spectral parameter imaging for detection of prognostically significant histologic features in uveal melanoma. Ultrasound Med Biol. 2003 Jul;29(7):951-9. doi: 10.1016/s0301-5629(03)00907-4. PMID 12878240
- [Result] Coleman DJ, Fish SK. Presbyopia, accommodation, and the mature catenary. Ophthalmology. 2001 Sep;108(9):1544-51. doi: 10.1016/s0161-6420(01)00691-1. PMID 11535447
- [Result] Silverman RH, Lizzi FL, Ursea BG, Rondeau MJ, Eldeen NB, Kaliscz A, Lloyd HO, Coleman DJ. High-resolution ultrasonic imaging and characterization of the ciliary body. Invest Ophthalmol Vis Sci. 2001 Apr;42(5):885-94. PMID 11274063
- [Result] Reinstein DZ, Silverman RH, Raevsky T, Simoni GJ, Lloyd HO, Najafi DJ, Rondeau MJ, Coleman DJ. Arc-scanning very high-frequency digital ultrasound for 3D pachymetric mapping of the corneal epithelium and stroma in laser in situ keratomileusis. J Refract Surg. 2000 Jul-Aug;16(4):414-30. doi: 10.3928/1081-597X-20000701-04. PMID 10939721
- [Result] Reinstein DZ, Silverman RH, Sutton HF, Coleman DJ. Very high-frequency ultrasound corneal analysis identifies anatomic correlates of optical complications of lamellar refractive surgery: anatomic diagnosis in lamellar surgery. Ophthalmology. 1999 Mar;106(3):474-82. doi: 10.1016/S0161-6420(99)90105-7. PMID 10080202
- [Result] Coleman DJ, Silverman RH, Daly SM, Rondeau MJ. Advances in ophthalmic ultrasound. Radiol Clin North Am. 1998 Nov;36(6):1073-82, x. doi: 10.1016/s0033-8389(05)70232-3. PMID 9884689
- [Result] Patel S, Reinstein DZ, Silverman RH, Coleman DJ. The shape of Bowman's layer in the human cornea. J Refract Surg. 1998 Nov-Dec;14(6):636-40. doi: 10.3928/1081-597X-19981101-11. PMID 9866103
- [Result] Kim DY, Reinstein DZ, Silverman RH, Najafi DJ, Belmont SC, Hatsis AP, Rozakis GW, Coleman DJ. Very high frequency ultrasound analysis of a new phakic posterior chamber intraocular lens in situ. Am J Ophthalmol. 1998 May;125(5):725-9. doi: 10.1016/s0002-9394(98)00025-7. PMID 9625568
- [Result] Ursea R, Coleman DJ, Silverman RH, Lizzi FL, Daly SM, Harrison W. Correlation of high-frequency ultrasound backscatter with tumor microstructure in iris melanoma. Ophthalmology. 1998 May;105(5):906-12. doi: 10.1016/S0161-6420(98)95036-9. PMID 9593396
- [Result] Cusumano A, Coleman DJ, Silverman RH, Reinstein DZ, Rondeau MJ, Ursea R, Daly SM, Lloyd HO. Three-dimensional ultrasound imaging. Clinical applications. Ophthalmology. 1998 Feb;105(2):300-6. doi: 10.1016/s0161-6420(98)93211-0. PMID 9479291
- [Result] Silverman RH, Folberg R, Boldt HC, Lloyd HO, Rondeau MJ, Mehaffey MG, Lizzi FL, Coleman DJ. Correlation of ultrasound parameter imaging with microcirculatory patterns in uveal melanomas. Ultrasound Med Biol. 1997;23(4):573-81. doi: 10.1016/s0301-5629(97)00037-9. PMID 9232766
- [Result] Silverman RH, Reinstein DZ, Raevsky T, Coleman DJ. Improved system for sonographic imaging and biometry of the cornea. J Ultrasound Med. 1997 Feb;16(2):117-24. doi: 10.7863/jum.1997.16.2.117. PMID 9166804
- [Result] Ursea R, Heinemann MH, Silverman RH, Deangelis LM, Daly SW, Coleman DJ. Ophthalmic, ultrasonographic findings in primary central nervous system lymphoma with ocular involvement. Retina. 1997;17(2):118-23. doi: 10.1097/00006982-199703000-00006. PMID 9143039
- [Result] Danias J, Aslanides IM, Eichenbaum JW, Silverman RH, Reinstein DZ, Coleman DJ. Iridoschisis: high frequency ultrasound imaging. Evidence for a genetic defect? Br J Ophthalmol. 1996 Dec;80(12):1063-7. doi: 10.1136/bjo.80.12.1063. PMID 9059271
- See also: Weill Cornell Ophthalmology Research — http://weillcornelleye.org/research/